CLINICAL TRIAL: NCT05653557
Title: Efficacy and Safety of Shen Que (RN8) Moxibustion on Reproductive Outcomes in Women of Advanced Reproductive Age (≥35 Years Old) With Unexpected Ovarian Poor Ovarian Response Undergoing in Vitro Fertilization and Embryo Transfer (IVF-ET): a Randomized Controlled Trial
Brief Title: Efficacy and Safety of Shen Que (RN8) Moxibustion in Unexpected POR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shandong University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Jing-Yan Song, Clinical Professor, Shandong University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SDUTCMSQPOR0113
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2024-01-09 (Actual); Status verified 2024-01

CONDITIONS: Infertility
Keywords: Shen Que (RN8); Moxibustion; In Vitro Fertilization and Embryo Transfer (IVF-ET); Poor Ovarian Response (POR); Poseidon Criteria
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Shen Que Moxibustion group (Experimental)
  Interventions: Other: Shen Que Moxibustion
- Control group (No Intervention)

INTERVENTIONS:
Other: Shen Que Moxibustion — Herb-partitioned moxibustion was administered at RN8 (Shen Que), once every 72 hours from the beginning of previous menstrual cycle day 2 until oocyte retrieval. Approximately 10 moxa cones will be used for this procedure, which will take approximately two hours. It is recommended that patients close their eyes during the procedure and rest. Following moxibustion, the umbilicus will be affixed and sealed with a medical applicator and removed after 24 hours.
  Arms: Shen Que Moxibustion group

SUMMARY:
Moxibustion of Shen Que (RN8) can increase the number of embryos available for transfer, thus improving pregnancy outcomes in women of advanced reproductive age who experience unexpected poor ovarian response.

DETAILED DESCRIPTION:
According to the traditional Chinese medicine (TCM) theory, Shen Que (RN8) is the place where the vitality converges under the navel, and is closely connected with the vitality generated by the kidney Qi. Therefore, stimulating Shen Que may stimulate the essence stored in the kidney, and improve the fertility of "五七" (≥ 35 years old) women.

Shen Que moxibustion has been shown to improve ovarian functional reserve in patients with ovarian insufficiency in previous studies. Nevertheless, studies on Shen Que moxibustion in advanced women with unexpected poor ovarian response (POR) who undergo IVF-ET are very limited. Consequently, we designed this randomized controlled trial to validate the hypothesis that Shen Que moxibustion improves reproductive outcomes in unexpected POR women.

ELIGIBILITY:
Inclusion Criteria:

* ≥35 years old with normal pre-stimulation ovarian reserve parameters (antral follicle count (AFC) ≥ 5 or anti-mullerian hormone (AMH) ≥1.2 ng/ml) and with an expected poor ovarian response (fewer than 4 oocytes) after standard ovarian stimulation.

Exclusion Criteria:

* Individuals with a Body Mass Index (BMI) ≥ 35 Kg/m2
* Those using the natural cycle or mild stimulation for IVF/intracytoplasmic sperm injection (ICSI) treatment
* Those with a history of unilateral oophorectomy or recurrent pregnancy loss, defined as two or more spontaneous abortions
* Acceptors of donated oocytes or performed either In vitro Maturation (IVM) or blastocyst biopsy for Preimplantation Genetic Diagnosis (PGD) or Preimplantation Genetic Testing for Aneuploidies (PGT-A)
* Those previously diagnosed with congenital (e.g., mediastinal uterus and double uterus) or acquired (e.g., submucosal myoma and adenomyosis) uterine abnormalities
* Patients with extremely advanced age ( ≥ 45 years old)
* Presence of a non-surgically treated hydrosalpinx or endometrial polyp and an ovarian endometriosis cyst requiring surgery, during ovarian stimulation

Ages: 35 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-12-15 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | One month
  Number of oocytes retrieved

SECONDARY OUTCOMES:
Cycle cancellation rate | One month
  Cycle cancellation is defined as cycle cancelled before obtaining at least one viable embryo for any reason. And cycle cancellation rate is calculated by dividing the number of women cancelled their cycle before obtaining at least one viable embryo for any reason by the total number of women randomized to the specific group.
Number of Metaphase II (MII) eggs | One month
  MII eggs is defined as eggs retrieved that reach the MII phase.
Cumulative Clinical pregnancy rate | Fourteen months
  Clinic pregnancy will be diagnosed with the detection of an intrauterine gestation sac. And cumulative clinic pregnancy rate is calculated by the number of women who achieves clinical pregnancy after transfers of all study-specific embryos (within 1 year after randomization) by the total number of women randomized to the specific group.
Implantation rate | Fourteen months
  Number of gestation sac detected / number of embryo transferred.
Good quality embryo rate | One month
  Good quality embryo is defined as embryo that is graded as 6-cell grade 2 (6CII) or better or blastocyst. And good quality embryo rate is calculated by dividing the number of good quality embryo by the total number of embryo obtained after fertilization in the specific group.
Cumulative live birth rate | Eighteen months
  Cumulative live birth rates (CLBR), defined as the proportion of deliveries with at least one live birth per started cycle or per oocyte aspiration, including all fresh and/or frozen embryo transfers until one delivery with a live birth or until all embryos were used.

CONTACTS AND LOCATIONS:
Locations (1):
- The Affiliated Hospital of Shandong University of Traditional Chinese Medicine, Jinan, Shandong, China

REFERENCES:
- [Derived] Song JY, Sun ZG, Ma YX. Efficacy and safety of Shen Que (RN8) moxibustion on reproductive outcomes in unexpected poor ovarian responders: a randomized controlled trial. J Ovarian Res. 2024 Aug 29;17(1):177. doi: 10.1186/s13048-024-01493-2. PMID 39210342